CLINICAL TRIAL: NCT05408247
Title: A Randomised Controlled Trial of N-acetylcysteine for the Management of Alcohol Use Disorder
Acronym: NAC-AUD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X21-0342
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: N-acetyl Cysteine; NAC; Alcohol Dependence; N-acetylcysteine
MeSH Terms: conditions — Alcoholism | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetyl Cysteine (Experimental): Generic name: N-acetyl cysteine. Brand: ACC-600 (Acetylcysteine). Strength: 600mg per capsule. Form: capsule Route: oral Frequency: 2x capsules twice per day = total 4 capsules/day Duration: 12 weeks
  + Standard of Care: Medical Management.
  Interventions: Drug: N-acetyl cysteine
- Placebo (Placebo Comparator): Matched placebo
  Generic name: dicalcium phosphate Strength: 600mg per capsule Form: capsule Route: oral Frequency: 2x capsules twice per day = total 4 capsules/day Duration: 12 weeks.
  + Standard of Care: Medical Management.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetyl cysteine — 2400mg/day
  Other Names: NAC
  Arms: N-acetyl Cysteine
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
To explore the effectiveness of n-acetylcysteine in improving treatment outcomes for alcohol use disorder in a double-blind randomised placebo-controlled trial.

DETAILED DESCRIPTION:
Australia urgently requires new treatment strategies for the treatment of alcohol dependence. Although alcohol use disorders are a leading cause of preventable death in Australia, their treatment is generally not evidence based. The medications currently approved for use in Australia for the management of alcohol dependence have limited efficacy, and existing research does not address the heterogeneity of treatment response. Targeted personalised medicine addresses this heterogeneity with better medicine selection for patients based on their genotype and clinical comorbidities.

Following on from a recent pilot study conducted by CI Morley (NCT03879759), this project will evaluate the clinical efficacy and tolerability of NAC, relative to a placebo, in heavy drinkers. We hypothesise that NAC-treated participants will be better able to achieve a reduction in heavy drinking. We will utilise a double-blind, randomised, controlled design. A sample of 280 individuals will receive 12 weeks of treatment with NAC (2400 mg/day) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Use Disorder according to the DSM-V criteria
* A desire to reduce or stop drinking
* Consumed at least 21 standard drinks per week or 2 heavy drinking days per week (HDD: ≥ 5 standard drinks/day for men; ≥4 for women) in the month prior to screening
* Adequate cognition and English language skills to give valid consent and complete research interviews
* Stable housing
* Willingness to give written informed consent

Exclusion Criteria:

* Pregnancy or lactation (women will be advised to use reliable contraception during the trial and a pregnancy test will be performed were necessary)
* Concurrent use of any psychotropic medication other than antidepressants (provided these are taken at stable doses for at least two months)
* Any substance dependence other than nicotine
* Clinically unstable systemic medical (e.g. cancer, end stage liver disease: e.g. MELD score ≥ 10) or psychiatric disorder (e.g. active psychosis, borderline personality disorder, active suicide risk: e.g. MADRAS item 10 score of 6) that precludes trial participation
* Concurrent use of selenium, vitamin D or other anti-oxidants
* Any alcohol pharmacotherapy within the past month

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Heavy Drinking Days | 24 weeks
  Reduction in Heavy Drinking Days (HDD; defined as 4 or more drinks in a day for women and five or more drinks in a day for men). This will be measured by the Timeline Follow Back and corroborated with Phosphatidylethanol (PEth) levels

SECONDARY OUTCOMES:
Changes in Liver Function | 24 weeks
  Liver Function will be assessed through blood sample at baseline. We will measurement levels of enzyme gamma-glutamyl transferase (GGT), aspartate transaminase (AST), and alanine transaminase (ALT).
Absence of any HDD | 24 weeks
  Measured by Timeline Follow Back and corroborated with Phosphatidylethanol (PEth) levels

OTHER OUTCOMES:
Cost-Efficacy | 12 weeks
  Examine the cost-efficacy between NAC and placebo from both health sector and societal perspectives. Measured by Disability-Adjusted Life Years (DALYs)
Changes in Alcohol Craving | 24 weeks
  As measured by the Alcohol Craving Experience Questionnaire (ACEQ). Higher scores indicate more severe craving.
Mean alcohol consumption per drinking day | 24 weeks
  Measured by Timeline Follow Back and corroborated with Phosphatidylethanol (PEth) levels
Change in dependence Severity | 24 weeks
  Measured by the Alcohol Dependence Scale. The minimum score is 0 and the maximum score is 47. A higher score indicates more severe dependence.
Changes in Anxiety | 24 weeks
  Measured by cumulative scores on the DASS-21 Anxiety Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates more anxiety.
Changes in Depression | 24 weeks
  Measured by cumulative scores on the DASS-21 Depression Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates greater depression.
Changes in Stress | 24 weeks
  Measured by cumulative scores on the DASS-21 Stress Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates more stress.
Sleep Disturbances | 24 weeks
  As measured by the ISI (Insomnia Severity Index). This Index has a minimum score of 0 and a maximum score of 28. The higher the score indicates more severe insomnia.
Lifetime Consequences related to Drinking | Baseline
  To examine the adverse consequences a participant has experienced in their lifetime due to alcohol abuse in five areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal. This is measured using the Drinker Inventory of Consequences Lifetime Edition (DrInC-2L). Higher scores indicate more consequences.
Recent Consequences related to Drinking | 12 weeks
  To examine the adverse consequences a participant has experienced in the last 3 months due to alcohol abuse in five areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal. This is measured using the Drinker Inventory of Consequences Recent Edition (DrInC-2R). Higher scores indicate more consequences.
Changes in Consequences related to Drinking | 24 weeks
  To examine the change in adverse consequences a participant has experienced across the trial due to alcohol abuse in five areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal. This is measured by comparing the Drinker Inventory of Consequences Recent Edition (DrInC-2R) and the Drinker Inventory of Consequences Lifetime Edition (DrInC-2L). Higher scores indicate more consequences.
Drinking Dairy | 12 weeks
  Daily texts will be sent out to participants querying the amount of alcohol they have consumed. Participant responses to this will be recorded. This will be managed through SEMA software.
Nicotine Dependence | Baseline
  Measured by the Fagerstrom Test for Nicotine Dependence (FTND). This test has a minimum score of 0 and a maximum score of 10. Higher scores indicate a more intense physical dependence on nicotine.
Changes in Suicidal Ideation | 24 weeks
  As measured by the Suicidal Ideation Attributes Scale (SIDAS). This scale has a minimum score of 0 and a maximum score of 50. Higher scores indicate more severe suicidal thoughts.
Changes in Information Gathering ability | 24 weeks
  As measured by the Caravan Spotter task of the Cognitive Impulsivity Suite (CIS). This measures information gathering through a perceptual decision making task whereby the target is initially ambiguous but progressively becomes clearer.
Changes in Attentional Control | 24 weeks
  As measured by the Bounty Hunter task of the Cognitive Impulsivity Suite (CIS). This measures attentional control using a Go/No Go task.
Changes in Monitoring of Feedback | 24 weeks
  As measured by the Prospectors Gamble task of the Cognitive Impulsivity Suite (CIS). This involves a probabilistic reverse learning task to measure monitoring of feedback.
Irritability | Baseline
  As measured by the Brief Irritability Test (BITe). This test has a minimum score of 0 and a maximum score of 30. Higher scores indicate greater irritability.
Changes in Physical Activity | 24 weeks
  To assess an individuals' health based on the previous 7 days of physical activity. This is measured by the International Physical Activity Questionnaire (IPAQ-Long). We are interested in whether across treatment, answers to this questionnaire will change.
Changes in Quality of Life | 24 weeks
  To assess whether treatment can change quality of life as measured by the short form Health Survey (SF-36). This survey has 36 items that measure 8 domains of health, including: physical functioning, physical role limitations, bodily pain, general health perceptions, energy/vitality, social functioning, emotional role limitations and mental health. The scores are transformed to range from 0 (worst possible health) to 100 (best possible health).
Changes in Quality of Life | 24 weeks
  As measured by the EQ-5D-5L. This instrument measures 5 different domains of life including: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is assessed by one question. This instrument has a minimum score of 0 (worst possible health) and a maximum score of 1 (best possible health).
Changes in ability to inhibit prepotent responses | 24 weeks
  As measured by the Stroop Colour Word Test. This test measures ability to inhibit prepotent responses and processing speed. This is assessed through the time it takes for an individual to appropriately select an incongruent response. For example, selecting "black" for the word "black" that is coloured in "green". Higher scores indicate worse performance.
Changes in processing speed | 24 weeks
  As measured by the Trail Making Task (TMT). This test measures the ability to an individual to process visual stimuli, as measured in time. In the TMT Part A, individuals are instructed to draw a line between numbers, 1-2-3-4-5. Higher time indicates slower processing speed. In the TMT Part B individuals are instructed to switch between drawing lines between numbers and letters, for example 1-A-2-B-3-C. Higher time indicates worse processing speed and switching ability.
Changes in DSM-5 PTSD symptomology | 24 weeks
  As measured by the PCL-5. This self-report questionnaire lists 20-items that assess DSM-5 PTSD criteria. A higher score indicates greater severity
Changes in use of Health Services | 24 weeks
  As measured by the Brief Health Services Use Questionnaire. This questionnaire assesses Health Service Use across the last 3 months.
Hangover Diary | 12 weeks
  Daily texts will be sent out to participants querying the hangover symptoms they are experiencing, if any. Participant responses to this will be recorded. This will be managed through SEMA software.
Using Redox Markers to predict treatment response | Baseline
  We will use blood samples collected at baseline to measure redox markers (GPxBC, GSHBC). At the end of treatment we will see whether these markers are predictive of treatment response
Changes in Redox Markers | 12 weeks
  We will use blood samples collected at baseline and wk 12 to measure changes in redox markers (GPxBC, GSHBC)

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Drug Health Services, Royal Prince Alfred Hospital, Sydney, New South Wales
  - Cornwall Street Medical Centre (UQ Health Care), Annerley, Queensland
  - Turning Point, Richmond, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morley K, Arunogiri S, Connor JP, Clark PJ, Chatterton ML, Baillie A, Slade T, Berk M, Lubman D, Haber PS. N-acetyl cysteine for the treatment of alcohol use disorder: study protocol for a multi-site, double-blind randomised controlled trial (NAC-AUD study). BMJ Open. 2025 Sep 8;15(9):e091631. doi: 10.1136/bmjopen-2024-091631. PMID 40921646